CLINICAL TRIAL: NCT04268524
Title: Randomised, Open Label, Multicentre, Non-inferiority Clinical Trial for New Treatment Modalities for Cutaneous Leishmaniasis Caused by Leishmania Tropica, in Pakistan
Brief Title: Randomised Clinical Trial for New Treatment Modalities for Cutaneous Leishmaniasis Caused by Leishmania Tropica, in Pakistan
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL_RCT_MF_vs_TT_2020
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Old World Cutaneous Leishmaniasis
Keywords: miltefosine; Thermotherapy
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Hyperthermia | interventions — miltefosine; Hyperthermia, Induced

STUDY DESIGN:
Intervention Model Description: randomised control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- monotherapy miltefosine (Experimental): Miltefosine capsules (Impavido®) 2.5 mg/kg daily PO for 28 days <30 kg BW allometric miltefosine dose based on fat-free mass. (approx. 2.5 mg/kg); >30 - ≤44kg BW: 100 mg/day BID; ≥45kg BW 150mg TDS
  Interventions: Combination Product: drug: miltefosine with thermotherapy
- Thermotherapy (Experimental): Thermotherapy (ThermoMed 1.8 ®) 50°C for 30 seconds, 1 session
  Interventions: Combination Product: drug: miltefosine with thermotherapy
- Combination miltefosine and thermotherapy (Experimental): Miltefosine capsules 2.5 mg/kg daily PO for 21days, and thermotherapy 50°C for 30 seconds, one session on day 1 of the miltefosine.
  Interventions: Combination Product: drug: miltefosine with thermotherapy
- ° Meglumine antimoniate (Glucantime®) intralesional (Active Comparator): Meglumine antimoniate (Glucantime®) intralesional injections 0.5-3ml, 8 sessions, bi-weekly

INTERVENTIONS:
Combination Product: drug: miltefosine with thermotherapy — see previous
  Other Names: device ThermoMed 1.8
  Arms: Combination miltefosine and thermotherapy; Thermotherapy; monotherapy miltefosine

SUMMARY:
randomised control clinical trial to evaluate miltefosine, thermotherapy and the combination miltefosine-thermotherapy are effective, safe and tolerable alternative treatment options to treat cutaneous leishmaniasis caused by L. tropica, in Pakistan compared to the standard of care.

DETAILED DESCRIPTION:
Until now, there is no well-established evidence based option to treat CL caused by the Leishmania tropica, besides antimonial injections. Alternative treatment options are not available in Pakistan, or there is limited evidence of the effectivity.

Effectiveness of thermotherapy in L. tropica is studied in only three studies in OWCL with a variable cure rate (54.1% - 98%). But it could be an attractive option, because only one treatment session is required and studies report less scarring tissue. Another promising treatment option is oral miltefosine. There is considerable evidence in the literature of the efficacy of miltefosine in treatment of CL caused by L. major, however no studies have been conducted to evaluate the efficacy in CL caused by L. tropica species. This oral treatment could have major benefits for CL patients as it can be provided in peripheral health facilities and to patients who have contraindications to antimony treatment (elderly, and patients with cardiac or renal disease, or diabetes). A combination of thermotherapy and miltefosine, the advantages offered by this combination are that a) the use of a topical plus a systemic treatment would hypothetically have an additive effect of two treatments with different modes of action. For the reason that systemic treatment could eliminate those circulating or remaining parasites located in the periphery of the lesion that topical treatment fails to remove, which might be the cause of a relapse, b) it may reduce the necessary length of treatment with miltefosine. For these above reasons, in a prospective trial we aim to evaluate the effectiveness and safety of thermotherapy, miltefosine and the combination of thermotherapy and miltefosine in CL caused by L. tropica, with the objective to find a treatment with an efficacy which is non-inferior to the standard of care with antimony injections.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with clinical and laboratory confirmed CL, and who can be treated with localised intralesional antimonial injections and/or thermotherapy:
* lesion size ≥0.5 cm and ≤4 cm
* not located on the ear, nose, near to the eye or mucosal membranes, on joints, or on a location that in the opinion of the principle investigator (PI) is difficult to apply thermotherapy (TT) or intralesional (IL) injections
* patient with ≤4 lesions
* duration of lesions less than five months by patient history
* Patients who have signed the informed consent form.

Exclusion Criteria:

* Pregnant women and breast feeding women
* Non-pregnant women in reproductive age refusing effective (injectable) contraception for a period of five months
* Patients <10years old
* Patients who cannot be treated with localised IL antimonial injections or TT (patients with more than 4 lesions, lesions >4cm in diameter, or located on joints, lips, nose, ears or near eyes)
* History of clinically significant medical problems or treatment that might interact with the study treatment and interact with wound healing, such as diabetes, vascular diseases and any immunocompromising condition
* Within eight weeks of trial D1 received treatment for leishmaniasis with any medication
* History of known or suspected hypersensitivity of idiosyncratic reactions to trial medication or excipients
* Has laboratory values at screening: serum creatinine above normal level; ALT 3 times above normal range
* Patient who is not willing to attend the trial visits, or is not able to comply with follow-up visits up to three months.
* Known history of drug addiction and/or alcohol abuse

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 832 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The initial clinical cure rate in each study arm | by Day 91.
  Initial Cure: Ulcerated lesions: 100% re-epithelialization of the lesion(s) Non-Ulcerated lesions: flattening and/or no signs of induration of the lesion(s) by Day 91.
Adverse events | by Day 91.
  Frequency, severity and seriousness of AEs by treatment group

SECONDARY OUTCOMES:
initial cure and no relapse | initial cure at D91 and have no relapse by D120.
  The proportion of patients in each study arm who have fulfilled the criteria of initial cure and have no relapse
100% re-epithelialized/ flattened | at visit until D120
  The number of patients with lesions 100% re-epithelialized/ flattened at each measurement time point.

CONTACTS AND LOCATIONS:
Overall Officials: Koert Ritmeijer, Study Director — Medecins Sans Frontieres, Netherlands
Locations (2):
- Pakistan (2):
  - Kuchlak Primary Health Care Centre (MCH), Kuchlagh, Balochistan
  - Shaheed Mohtarma Benazir Bhutto General Hospital, Quetta, Balochistan

IPD SHARING:
Plan to Share IPD: Undecided
Plan need to be made what wilkl be shared with whom (such as study protocol, SAP, ICF etc)